CLINICAL TRIAL: NCT04801966
Title: Safety and Oversight of the Individually Tailored Treatment Approach: A Novel Pilot Study
Acronym: TAILOR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20/029
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — trametinib; cobimetinib; binimetinib; Alpelisib; Vemurafenib; dabrafenib; encorafenib; palbociclib; olaparib; ribociclib; abemaciclib; talazoparib; Nivolumab; atezolizumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): All participants will have an individualised treatment plan. The possible treatments that can be prescribed are as follows, they may be given as a single agent or in combination
  * Trametinib 2 mg/day
  * Cobimetinib 60 mg/day, on day 1-21 of each 28 day cycle (21 days on, 7 days off)
  * Binimetinib 45 mg/ twice a day
  * Alpelisib 300 mg/day
  * Vemurafenib 960 mg twice a day
  * Dabrafenib 150 mg twice a day
  * Encorafenib 450 mg/day
  * Palbociclib 125 mg/day, on day 1-21 of each 28 day cycle (21 days on, 7 days off)
  * Ribociclib 600 mg/day, on day 1-21 of each 28 day cycle (21 days on, 7 days off
  * Abemaciclib 150 mg twice a day
  * Olaparib 300 mg twice a day
  * Talazoparib 1 mg/day
  * Nivolumab 240 mg IV once every two weeks
  * Atezolizumab 1200 mg IV on day 1 of a 21 day cycle
  * Pembrolizumab 200 mg IV on day 1 of a 21 day cycle
  Interventions: Drug: Trametinib; Drug: Cobimetinib; Drug: Binimetinib; Drug: Alpelisib; Drug: Vemurafenib; Drug: Dabrafenib; Drug: Encorafenib; Drug: Palbociclib; Drug: Olaparib; Drug: Ribociclib; Drug: Abemaciclib; Drug: Talazoparib; Drug: Nivolumab; Drug: Atezolizumab; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Trametinib — 2 mg per day, continuous
Drug: Cobimetinib — 60 mg/day for 21 days of a 28 day cycle
Drug: Binimetinib — 45 mg/twice a day, continuous
Drug: Alpelisib — 300 mg/day, continuous
Drug: Vemurafenib — 960 mg/twice per day, continuous
Drug: Dabrafenib — 150 mg/twicce per day, continuous
Drug: Encorafenib — 450 mg/day, continuous
Drug: Palbociclib — 125 mg/day, day 1-21 of a 28 day cycle
Drug: Olaparib — 300 mg/twice per day, continuous
Drug: Ribociclib — 600 mg/day, on day 1 -21 of a 28 day cycle
Drug: Abemaciclib — 150 mg twice/day, continuous
Drug: Talazoparib — 1 mg/day, on day 1 -28 of each 28 day cycle
Drug: Nivolumab — 240 mg IV once every 2 weeks
Drug: Atezolizumab — 1200 mg IV on Day 1 of a 21 day cycle
Drug: Pembrolizumab — 200 mg IV on day 1 of a 21 day cycle

SUMMARY:
This study is looking at outcomes in people with advanced cancers who have exhausted standard treatment options and are accessing off indication or unregistered drugs or combinations of drugs through compassionate access from the manufacturer.

DETAILED DESCRIPTION:
Some advanced cancers have numerous standard treatment options that have proven efficacy in clinical trials. However, in other cancers, there may be few or no standard treatment options with proven efficacy as determined in a large clinical trial. This may be particularly the case for rare cancers in which there is a lack of clinical research. When seriously ill patients run out of standard treatment options, they will often consider non-standard treatment options (such as treatments that are currently unapproved by the regulatory agency for the given indication). The majority of clinicians and researchers agree that this is best received in a clinical trial setting as this provides ethical and clinical oversight, as well as addresses prospectively defined research questions which can be publicly reported. This allows the conclusions of the research to be available to the entire clinical and research community.

In general, an access program enables patient access to a non-reimbursed therapeutic agent, outside of a clinical trial setting. Compassionate access is typically for therapeutics that are not yet approved or TGA registered, and are still considered investigational. In general, there is a negotiation between the pharmaceutical company and the clinician and patient regarding access to the therapeutic agent, as well as whether the medicine will be provided free of charge, or on some form of cost-sharing arrangement. In Australia, access to TGA non-registered medicines also requires an application via the "Special Access Scheme". For most cancer patients, the use falls under category A, for a patient defined as seriously ill. This sub-study generally pertains to compassionate access to therapeutic agents. Given the ad hoc nature of compassionate access for patients, there is relatively little reported data on clinical outcomes.

Compassionate access is an established process with increasing demands. This study is designed to provide a framework for which patients treated with compassionate access therapeutics can register, so that some of the limitations of ad hoc compassionate access programs can be overcome.

A study committee will prospectively assess each individual patient's detailed treatment approach in an objective and time-efficient manner. If approved, the patient may be eligible to register into the treatment phase of the study. The study committee is essential to provide a balanced approach to understanding the rationale for the study treatment, as well as potential safety issues that may arise. As previously reported, this is an essential component to improving patient oversight as well as equity

ELIGIBILITY:
Inclusion Criteria:

1. Patient or their parent(s)/legal guardian(s) has provided written informed consent using the main study PICF
2. Continues to meet all the inclusion criteria as per the TRIAGE Framework protocol as follows:

   1. Male or female patient, aged 2 years or older
   2. Patient has pathologically confirmed locally advanced, incurable or metastatic cancer of any histological type
   3. Have an available TRIAGE sub-study with a matched therapy
   4. Documented progression following standard therapy, or for whom, in the opinion of the Investigator, no appropriate standard therapy exists
   5. Life expectancy of > 3 months
   6. Adequate performance status:

   i. For patients aged 18 years or over, Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (appendix 1) ii. For patients aged 17 years, Karnofsky score ≥ 50 (appendix 2) iii. For patients aged 16 years or under, Lansky score ≥ 50 (appendix 3)
3. Treatment regimen and schedule of assessments that has been approved by the TAILOR Study Committee
4. Approved treatment is obtainable
5. Patient has measurable disease or evaluable disease as defined by RECIST 1.1 (or RANO criteria for primary CNS cancers or the Cheson (IWG) revised response criteria for lymphomas)
6. Patient must have adequate bone marrow, hepatic and renal function within 7 days prior to registration:

   * ANC ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L (platelet count ≥ 50 x 109/L for haematological malignancy indications)
   * ALT ≤ 2.5x ULN, unless liver metastases or invasion are present, in which case it must be ≤ 5x ULN
   * AST ≤ 2.5x ULN, unless liver metastases or invasion are present, in which case it must be ≤ 5x ULN
   * Total bilirubin ≤ 1.5x ULN except patients with Gilbert's Syndrome, who are eligible in consultation with their physician
   * Serum creatinine ≤ 1.5x ULN
7. Patient is willing and able to comply with the protocol for the duration of the study including undergoing, treatment, and scheduled visits and examination including follow up
8. Female patients of childbearing potential must have a negative serum pregnancy test at screening for the main study and agree to use highly effective methods of birth control while receiving approved treatment through to the time frame specified in the approved ITAP after the last dose. Patients of childbearing potential are those who have not been surgically sterilised or have not been free from menses for > 1 year.
9. Sexually active males must agree to use a condom during intercourse while taking the approved treatment through to the time frame specified in the approved ITAP after the last dose and should not father a child in this period.

Exclusion Criteria:

1. One or more of the exclusion criteria as per the TRIAGE Framework protocol applies as follows:

   1. Significant cardiovascular disease
   2. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
   3. Other co-morbidities or conditions that may compromise assessment of key outcomes or in the opinion of the clinician, limit the ability of the patient to comply with the protocol
2. Any unresolved toxicity (≥CTCAE grade 2) from previous anti-cancer therapy, with the exception of alopecia.

   Patients with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product(s) may be included (e.g. hearing loss, peripheral neuropathy)
3. Symptomatic, or actively progressing CNS metastases (unless a primary brain tumour).Patients with a history of treated

   CNS lesions are eligible, provided that all of the following criteria are met:

   Measurable disease per RECIST 1.1 must be present outside the CNS Metastases are limited to the cerebellum or the supratentorial region (i.e. no metastases to the midbrain, pons, medulla, or spinal cord) There is no clinical evidence of interim progression between completion of CNS-directed therapy and registration on the study (radiological re-assessment is not required) The patient has not received radiotherapy within 14 days prior to registration Anticonvulsant therapy at a stable dose is permitted
4. History of leptomeningeal disease unless a primary brain tumour
5. Known active infection including tuberculosis, HBV, HCV, or HIV. Patients with a past or resolved HBV infection (defined as the presence of HBcAb and absence of HBsAg) are eligible. Patients with a past or resolved HCV infection are eligible only if polymerase chain reaction is negative for HCV RNA

Additional inclusion and/or exclusion criteria for the main study will be stipulated in the approved Individualised Treatment and Assessment Plan as each treatment regimen is expected to have specific requirements.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Safety of the study design as mechanism for administering individualised therapies to individuals with incurable malignancies | At the end of the study, approximately 5 years after the first participant commences treatment
  Severity of adverse events as determined by NCI CTCAE v5.0
Feasibility of the study design as mechanism for administering individualised therapies to individuals with incurable malignancies | At the end of the study, approximately 5 years after the first participant commences treatment
  Feasibility measured by:
  Number of treatment plans proposed to the study committee Proportion of treatment plans proposed that are approved Proportion of approved plans for which study drug(s) were obtained Proportion of approved plans for which study drug(s) were obtained and patient was registered on the trial

SECONDARY OUTCOMES:
Efficacy of individualised therapies in patients registered to the study | At the end of the study, approximately 5 years after the first participant commences treatment
  Efficacy measured by:
  * Objective response rate (ORR), defined as the proportion of patients with an objective response (partial response [PR] or complete response [CR]), as determined by the Investigator by RECIST 1.1 (or RANO for primary CNS cancers or Cheson IWG for lymphomas)
  * Clinical benefit rate (CBR), defined as the proportion of patients with CR, PR, or stable disease for ≥ 4 months, as determined by the Investigator by RECIST 1.1 (or RANO for primary CNS cancers or Cheson IWG for lymphomas)
  * Progression-free survival (PFS), defined as the time from registration to the first occurrence of disease progression, as determined by the Investigator according to RECIST 1.1 or RANO for primary CNS cancers or Cheson IWG for lymphomas, or death from any cause, whichever occurs first.
  * Overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Luen, MBBS, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
The Sponsor will consider individual requests to share data